CLINICAL TRIAL: NCT06572163
Title: Clinical Validation Study of the Eximis CS (Contained Segmentation) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eximis Surgical (Industry)
Collaborators: Proxima CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP2024-001
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Laparoscopic Gynecological Surgical Procedures
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surgical (Other): containment, segmentation, and extraction of uterine tissue
  Interventions: Device: Eximis CS (Contained Segmentation) System

INTERVENTIONS:
Device: Eximis CS (Contained Segmentation) System — The Eximis CS System is an integrated system consisting of a 900 mL Capture Bag, Inflation Mechanism, two Eximis Segmenters, and the Eximis RF Generator.

SUMMARY:
The purpose of this study is to evaluate device safety and effectiveness of the Eximis CS System.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to confirm device safety and effectiveness when utilized for containment, segmentation, and extraction of uterine tissue in pre-menopausal women undergoing laparoscopic hysterectomy or myomectomy for non-cancer indications.

Eligible subjects who have signed an informed consent form (ICF) will be enrolled. Subjects will be sequentially enrolled and assigned a study identification number. Surgeons will also be assigned a unique number.

Subjects will undergo the standard of care regarding all aspects of the pre-operative, surgical, and follow-up procedures. The aspect unique to this study is the capture, segmentation, and extraction of the target tissue will utilize one integrated device, the Eximis CS System, which segments tissue via segmenting wires using RF energy. The device is not intended to provide any therapeutic effect.

All subjects will be followed for safety through two post-procedure follow-up visits. One will be scheduled at a minimum of 14 days and a maximum of 21 days post-operatively. The second will be a follow-up phone call scheduled at a minimum of 30 days and a maximum of 45 days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

Planned laparoscopic hysterectomy or myomectomy. Tissue specimen size is greater than 6 cm in diameter, less than 13 cm in the longest dimension, and at most 10 cm in the second longest dimension, based on preoperative assessment.

Pre-operative evaluation, which may include imaging, cervical cancer screening, and endometrial biopsy has been completed.

Signed informed consent. Willing to adhere to protocol requirements and complete follow-up.

Exclusion Criteria:

Subject is post-menopausal, defined as amenorrhea >12 months in the absence of ovulation suppression.

Known or suspected malignancy of gynecological origin as determined by standard clinical practice.

Candidate for en bloc tissue removal, for example through the vagina or via a mini-laparotomy incision.

Hemoglobin < 8 g/dl within 30 days prior to surgery. Subject has a current history of undiagnosed genital bleeding Subject has an implanted electronic device where use of radiofrequency (RF) energy would be contraindicated (e.g., pacemaker, internal defibrillator).

Medical condition, surgical history, or intra-operative findings, which in the option of the investigator, precludes utilization of the Eximis CS System.

Known allergy to polyurethane, polyethylene, thermoplastic fluoropolymer and/or chlorinated polyvinyl chloride.

Concurrent participation in another therapeutic or interventional clinical trial with investigational pharmaceutical agent(s) or medical device(s) that could impact evaluation of this study as determined by the Investigator.

Inability to comply with the study procedures or follow-up in the opinion of the investigator.

Subject is pregnant.

Intraoperative Exclusion: Abdominal wall thickness at the umbilicus incision site exceeds 6 cm.

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
Performance | 2 months
  Percentage of procedures successfully completed with use of the Eximis CS device per the Instructions for Use and without breach of the containment bag.

SECONDARY OUTCOMES:
Usability | 2 months
  Percentage of procedures where all critical tasks related to the Eximis CS are performed without observed failure or omission.
  Percentage of procedures requiring critical troubleshooting steps (i.e., extending an incision, employing alternate tissue removal techniques) per the Instructions for Use Percentage of procedures requiring other troubleshooting steps (i.e., replacing the RF Generator, Segmenter, or Capture Bag; cutting Segmenter wires; responding to an alarm or information signal) per the Instructions for Use

OTHER OUTCOMES:
Adverse Events | 2 months
  The incidence of device-related adverse events. The incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Unanticipated Adverse Device Effects (UADEs)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Chudnoff, MD, Principal Investigator — Maimonides Medical Center
Locations (4):
- United States (4):
  - Advent Health, 410 Celebration Place, Celebration, Florida
  - Rosemark Womens Care Specialists, Idaho Falls, Idaho
  - Maimonides Medical Center, Brooklyn, New York
  - Oregon Health and Science University School of Medicine, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided